CLINICAL TRIAL: NCT00032188
Title: A Randomized Phase II Study Of Interluekin-2 In Combination With Three Different Doses Of Bryostatin In Patients With Renal Cell Carcinoma
Brief Title: Interleukin-2 and Bryostatin 1 in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02460; 11367; N01CM17102 (NIH); CDR0000069267 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — aldesleukin; Interleukin-2; bryostatin 1; Bryostatins

ARMS (3):
- Arm I (aldesleukin and lowest dose bryostatin 1) (Experimental): Patients receive IL-2 subcutaneously on days 1-4, 8-11, and 15-18. For the second and subsequent courses of IL-2, patients also receive lowest dose bryostatin 1 IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: aldesleukin; Drug: bryostatin 1; Other: laboratory biomarker analysis
- Arm II (aldesleukin and middle dose bryostatin 1) (Experimental): Patients receive IL-2 subcutaneously on days 1-4, 8-11, and 15-18. For the second and subsequent courses of IL-2, patients also receive middle dose bryostatin 1 IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: aldesleukin; Drug: bryostatin 1; Other: laboratory biomarker analysis
- Arm III (aldesleukin and highest dose bryostatin 1) (Experimental): Patients receive IL-2 subcutaneously on days 1-4, 8-11, and 15-18. For the second and subsequent courses of IL-2, patients also receive highest dose bryostatin 1 IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: aldesleukin; Drug: bryostatin 1; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: aldesleukin — Given subcutaneously
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Drug: bryostatin 1 — Given IV
  Other Names: B705008K112; BRYO; Bryostatin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining bryostatin 1 with interleukin-2 may cause a stronger immune response and kill more tumor cells. Randomized phase II trial to study the effectiveness of combining interleukin-2 and bryostatin 1 in treating patients who have advanced kidney cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with advanced renal cell carcinoma treated with interleukin-2 (IL-2) and bryostatin 1.

II. Compare the toxicity of 3 different doses of bryostatin 1 given in combination with a fixed dose of IL-2 in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of three dose levels of bryostatin 1.

ARM I: Patients receive interleukin-2 (IL-2) subcutaneously on days 1-4, 8-11, and 15-18. For the second and subsequent courses of IL-2, patients also receive lowest dose bryostatin 1 IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive IL-2 as in arm I and middle dose bryostatin 1 IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive IL-2 as in arm I and highest dose bryostatin 1 IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

Patients with stable or responding disease may receive 3 additional courses of therapy. An additional cohort of patients receives treatment as above at a higher dose to evaluate toxicity.

Patients are followed for 1 year.

PROJECTED ACCRUAL: A total of 24-65 patients (8-16 per bryostatin 1 dose level) will be accrued for this study within 14-27 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell carcinoma

  * Recurrent or refractory advanced disease
  * Newly diagnosed disease with no appropriate standard therapy available
* Measurable disease
* No active CNS metastases

  * Single prior CNS metastasis allowed if all of the following are true:

    * Previously resected and irradiated
    * No evidence of progressive CNS disease for at least 8 weeks after completion of therapy
    * No requirement for steroids or anti-seizure medications
* Performance status - ECOG 0-2
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN
* Creatinine no greater than 2.0 mg/dL
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 2 weeks after study for female patients and for 3 months after study for male patients
* No concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study entry
* No prior interleukin-2
* See Disease Characteristics
* See Disease Characteristics
* Prior radiotherapy to less than 50% of bone marrow allowed
* At least 4 weeks since prior radiotherapy
* See Disease Characteristics
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2002-01; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Overall response (CR and PR) | Up to 1 year
  Will be comparing using Fisher's exact test.
Time to disease progression | From the date of registration to the date of progressive disease or death
  Kaplan-Meier estimates will be generated.
Overall survival | Up to 1 year
  Kaplan-Meier estimates will be generated.
Disease-free survival | Up to 1 year
  Will be compared using the logrank test.

SECONDARY OUTCOMES:
All observed toxicities assessed using CTC version 2.0 | Up to 1 year
  A chi-square test and one-way ANOVA will be used for categorical and continuous toxicity endpoints, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States